CLINICAL TRIAL: NCT05908214
Title: The Application of Wide Pulse High Frequency Neuromuscular Electrical Stimulation in Disorders Associated With Motoneuron Hyperexcitability
Acronym: MnHyperex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Nicolas Place, Professor, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01817
Record Dates: First submitted 2023-05-16; First posted 2023-06-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Cramp; Restless Legs Syndrome; Healthy Volunteers
Keywords: muscle strength; persistent inward current; training
MeSH Terms: conditions — Stroke; Muscle Cramp; Restless Legs Syndrome

STUDY DESIGN:
Intervention Model Description: Stroke patients in the training group will be compared to stroke patients in the control group.
  Participants prone to cramps will be compared to healthy participants. Patients with restless legs syndrome will be compared to healthy participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke patients - training group (Experimental): Participants in this group will take part in a 6-week WPHF NMES training period and plantar flexor neuromuscular function will be assessed before and after training.
  Interventions: Other: wide pulse high frequency neuromuscular electrical stimulation training
- stroke patients - control group (No Intervention): Participants in this group will keep their daily life activities for 6 weeks and plantar flexor neuromuscular function will be assessed before and after training.

INTERVENTIONS:
Other: wide pulse high frequency neuromuscular electrical stimulation training — Plantar flexors will be stimulated with wide pulse high frequency neuromuscular electrical stimulation 3 times a week for 6 weeks
  Arms: Stroke patients - training group

SUMMARY:
In the present project, the investigators aim at proposing innovative ways of investigating spinal motoneuron hyperexcitability to counteract the associated impairments by using wide pulse high frequency neuromuscular electrical stimulation (WPHF NMES) in various populations. The investigators will use WPHF NMES contractions as a model to gain insights into the mechanisms underlying muscle cramps, restless legs syndrome or stroke-induced spasticity as there is evidence that they share common underlying mechanisms. The investigators will then use WPHF NMES as a training modality to improve plantar flexor neuromuscular function in stroke patients by taking advantage of their motoneuronal hyperexcitability.

ELIGIBILITY:
STROKE PATIENTS:

* Diagnosis of first-ever stroke (ischemic or hemorrhagic) with unilateral motor deficits from at least 6 months. Stroke will have to be confirmed from medical records and/or radiological imaging (CT scan or MRI)
* Inadequate ankle control during gait defined as ankle dorsiflexion less than 5° during stance phase and 0° during swing phase; 0° = ankle neutral position)
* Passive range of motion of ankle dorsiflexion at least to neutral position
* Ability to walk at least 10 m with or without assistive devices
* Spasticity at the triceps surae (either soleus and/or gastrocnemii) considered as a Modified Ashworth Sore ≥1
* Being available for the study period and willing to participate
* No contraindication to neuromuscular electrical stimulation

Contraindications for stroke patients:

* Surface sensory loss of affected lower leg (defined as incapacity to feel the 60-g touch using the Semmes-Weinstein monofilament test)
* Patients unable to understand indications or to provide informed consent
* A history of orthopedic or other neurological disorders affecting walking function
* A history of surgery to correct drop foot (ankle fixation)
* Patients under antispastic medication (baclofen, tizanidine, tolperisone, benzodiazepines, dantrolene or botulinum toxin to the plantar flexor muscles in the last 6 months).

PEOPLE PRONE TO MUSCLE CRAMPS:

* Reporting nocturnal muscle cramps (the assessment will be done through a questionnaire)
* Not being treated for muscle cramps
* Being available for the study period and willing to participate
* No contraindication to neuromuscular electrical stimulation

PATIENTS WITH RESTLESS LEGS SYNDROME:

To be included in the study, RLS patients will have to satisfy the Diagnostic criteria for RLS published by the International Restless Legs Syndrome StudyGroup (IRLSSG). All five key clinical features are required for the diagnosis:

* An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs. Sometimes the urge to move is present without the uncomfortable sensations, and sometimes the arms or other body parts are involved in addition to the legs.
* The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying or sitting.
* The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues.
* The urge to move or unpleasant sensations are worse in the evening or night than during the day, or only occur in the evening or night. When symptoms are severe, the worsening at night may not be noticeable but must have been previously present.
* Symptoms are not solely accounted for by another medical or behavioral condition, such as leg cramps or habitual foot tapping.
* No contraindication to neuromuscular electrical stimulation

They will also have to satisfy the following criteria:

* Diagnosis of primary RLS corresponding to:

  1. The presence of periodic limb movements
  2. A dopaminergic treatment response
  3. The presence of RLS in first-degree relatives
  4. A lack of profound daytime sleepiness
* Being available for the study period and willing to participate

HEALTHY PARTICIPANTS:

* No neurological disease
* No contraindication to neuromuscular electrical stimulation
* Being available for the study period and willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in maximal voluntary contraction force | through study completion, an average of 8 weeks
  Change from baseline maximal voluntary contraction force after the six-week training period in stroke patients
Change in NMES-evoked force | through study completion, an average of 8 weeks
  Change from baseline NMES-evoked force after the six-week training period
NMES-evoked force | through study completion, an average of 2 weeks
  Comparison of NMES-evoked force in plantar flexor muscles between patients (prone to cramps or restless legs) and healthy volunteers
Change in estimates of persistent inward current (Delta F assessed with high-density surface electromyography and/ or the torque measured during vibration after the last bout of NMES) | through study completion, an average of 8 weeks
  Change from baseline estimates of persistent inward current after the six-week training period in stroke patients
Estimates of persistent inward current (Delta F assessed with high-density surface electromyography and/ or the torque measured during vibration after the last bout of NMES) | through study completion, an average of 8 weeks
  comparison of estimates of persistent inward current strength in plantar flexor muscles between patients (prone to cramps or restless legs) and healthy volunteers

SECONDARY OUTCOMES:
Change in voluntary activation level and contractile properties of the plantar flexor muscles | through study completion, an average of 8 weeks
  Change from baseline voluntary activation level and contractile properties of the plantar flexor muscles after the six-week training period in stroke patients
voluntary activation level and contractile properties of the plantar flexor muscles | through study completion, an average of 2 weeks
  comparison of voluntary activation level and contractile properties of the plantar flexor muscles between patients (prone to cramps or restless legs) and healthy volunteers
change in spasticity at the ankle joint level for stroke patients | through study completion, an average of 8 weeks
  Change from baseline Ashworth scale score (minimal score 0, maximal score 4, a higher score means a worst outcome) after the six-week training period in stroke patients
10-m walking test (s) | through study completion, an average of 8 weeks
  functional test
6-min walking test (m) | through study completion, an average of 8 weeks
  functional test
time up and go test (s) | through study completion, an average of 8 weeks
  functional test
Change in spinal excitability in stroke patients | through study completion, an average of 8 weeks
  change from baseline soleus Hoffmann reflex amplitude after the six-week training period in stroke patients
Spinal excitability | through study completion, an average of 2 weeks
  comparison of soleus Hoffmann reflex amplitude between patients (prone to cramps or restless legs) and healthy volunteers
Cramp threshold frequency (CTF) for cramp-prone individuals | through study completion, an average of 2 weeks
  comparison between participants reporting muscle cramps and healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Bâtiment Synathlon, quartier UNIL-Centre, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided